CLINICAL TRIAL: NCT02385591
Title: Innovative Physical Activity Interventions for Overweight Latinos
Acronym: SMS-Stanford
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Abby C King, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DK102016 (NIH); R01DK102016 (NIH)
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Sedentary Lifestyle
Keywords: physical activity; Latinos; overweight; SMS; mHealth
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Telephone Support (Experimental): Participants will receive bi-weekly 20 minute telephone calls from a trained professional facilitator offering physical activity advice with the goal of increasing moderate-to-vigorous intensity physical activity.
  Interventions: Behavioral: Telephone Support
- SMS Support (Experimental): Participants will receive weekly text messages (3-5 text messages per week) offering physical activity advice with the aim of increasing moderate-to-vigorous intensity physical activity.
  Interventions: Behavioral: SMS Support
- Attention-control (Active Comparator): Participants will receive telephone-based general nutrition advice.
  Interventions: Behavioral: SMS Support

INTERVENTIONS:
Behavioral: Telephone Support — telephone-based physical activity advice and support delivered by a trained professional facilitator.
  Other Names: Active Choices
  Arms: Telephone Support
Behavioral: SMS Support — Telephone-based physical activity advice and support delivered by SMS.
  Arms: Attention-control; SMS Support

SUMMARY:
This research aims to investigate the effectiveness of an automated Simple Message Service (SMS, also known as text messaging) advisor system relative to a proven human advisor program to promote regular, sustained physical activity among inactive, overweight Latinos. The SMS Advisor program represents a potentially lower-cost and high yield alternative to person-delivered health promotion programs that could be more rapidly disseminated with greater and faster uptake.

DETAILED DESCRIPTION:
Latinos are the fastest growing ethnic group in the US and are disproportionately impacted by chronic conditions (e.g., overweight/obesity, diabetes) that can be mitigated by physical activity. While evidence-based programs are available to improve physical activity, dissemination is constrained by reliance on costly, limited resources. Short message service (SMS or text messaging) has strong potential as an intervention medium for Latinos, as they are dominant users of mobile phones and text messaging, including those with limited literacy and computer skills. The investigators propose to develop a personalized, culturally-congruent and interactive SMS program to promote the adoption and maintenance of physical activity for overweight, underactive Latino adults and test it for comparable efficacy to an evidence-based telephone-based advising program that has been used successfully with Latinos. Grounded in Social Cognitive and Self-Determination Theories, both programs will include a core set of self-regulatory skill building, social support, and autonomous motivation enhancement, and will be tailored for cultural, linguistic and literacy appropriateness. Randomized at the individual level, 376 sedentary, overweight Latinos ages 45 years and older will be assigned to one of three arms: the SMS-delivered physical activity program, the Human-delivered physical activity program, or an attention-control arm of SMS-delivered basic healthful nutrition advice. They will receive their assigned program for 12 months, and then will be followed for a 6-month maintenance phase, with a final assessment at 18 months. Analyses will determine if the two physical activity programs result in equivalent efficacy in adoption and maintenance of clinically meaningful physical activity increases, and superiority over the attention-control arm at 12 and 18 months. The two physical activity interventions will also be compared for equivalency in prevention of weight gain and reduction in abdominal adiposity. The investigators will explore the relative costs of the programs to determine which program increases physical activity for a lower cost. While health promotion programs delivered by professional staff may be more expensive than those delivered electronically, it is unclear if the automated version can produce more cost-efficient outcomes (i.e., comparable improvements in outcomes for significantly reduced cost). This study will determine if SMS is equivalent in efficacy to the traditional human-delivery channel in increasing physical activity and preventing weight gain, and if it results in a more cost-efficient program. If achieved, this research can significantly reduce health disparities associated with physical activity for Latinos by providing an efficacious, tailored and culturally appropriate program poised for widespread dissemination and rapid uptake.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified Latino ethnicity;
* Body Mass Index between 25 and 40;
* Aged greater than or equal to 35 years
* Physically inactive (i.e., not engaged in moderate- or greater intensity PA at least 60 minutes/week over the past 6 months);
* Stable on all medications over the past 3 months;
* Regular access to a mobile phone;
* Willing to accept random assignment, and willing to complete all assessments.

Exclusion Criteria:

* Aged less than 35 years
* Body Mass Index greater than 40
* Physically active (i.e., engaged in moderate- or greater intensity PA for more than 60 minutes/week over the past 6 months);
* Not stable on all medications over the past 3 months;
* No regular access to a mobile phone;
* Not willing to accept random assignment and/or willing to complete all assessments.
* Medical contraindications to regular unsupervised PA, including uncontrolled metabolic disorders;
* Unable to understand English or Spanish sufficiently to provide informed consent

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Change in weekly walking minutes from baseline to 12 months | baseline, 6 months, 12 months
  Total weekly walking minutes measured by CHAMPS questionnaire (Stewart AL, Mills KM, King AC, Haskell WL, Gillis D, Ritter PL. CHAMPS physical activity questionnaire for older adults: outcomes for interventions. Med Sci Sports Exerc. 2001 Jul;33(7):1126-41)

SECONDARY OUTCOMES:
Body weight stability from baseline to 12 months | baseline, 6 months, 12 months
  body weight measured by portable digital scale in kg
Change in moderate-to-vigorous physical activity from baseline to 12 months | baseline, 6 months, 12 months
  Moderate-to-vigorous physical activity measured by CHAMPS questionnaire (Stewart AL, Mills KM, King AC, Haskell WL, Gillis D, Ritter PL. CHAMPS physical activity questionnaire for older adults: outcomes for interventions. Med Sci Sports Exerc. 2001 Jul;33(7):1126-41)

CONTACTS AND LOCATIONS:
Overall Officials: Abby C King, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Prevention Research Center, Palo Alto, California, United States

REFERENCES:
- [Result] Stewart AL, Mills KM, King AC, Haskell WL, Gillis D, Ritter PL. CHAMPS physical activity questionnaire for older adults: outcomes for interventions. Med Sci Sports Exerc. 2001 Jul;33(7):1126-41. doi: 10.1097/00005768-200107000-00010. PMID 11445760
- [Derived] King AC, Campero MI, Rodriguez Espinosa P, Garcia D, Corral C, Sweet CC, Xiao L, Royer MF, Zamora A, Cortes AL, Done M, Banda JA. Human Telephone vs Text Message Counseling and Physical Activity Among Midlife and Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2528858. doi: 10.1001/jamanetworkopen.2025.28858. PMID 40906479
- [Derived] King AC, Campero I, Sheats JL, Castro Sweet CM, Espinosa PR, Garcia D, Hauser M, Done M, Patel ML, Parikh NM, Corral C, Ahn DK. Testing the effectiveness of physical activity advice delivered via text messaging vs. human phone advisors in a Latino population: The On The Move randomized controlled trial design and methods. Contemp Clin Trials. 2020 Aug;95:106084. doi: 10.1016/j.cct.2020.106084. Epub 2020 Jul 11. PMID 32659437